CLINICAL TRIAL: NCT04315623
Title: Regional Citrate Anticoagulation Versus No-anticoagulation for CRRT in Hyperlactatemia Patients With Increased Bleeding Risk: a Randomized, Control, Open-labeled Clinical Trial
Brief Title: RCA for CRRT in Hyperlactatemia Patient With Increased Bleeding Risk
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Air Force Military Medical University, China (Other)
Responsible Party: Principal Investigator, Shiren sun, Professor, Air Force Military Medical University, China
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RCA-CRRT-Hyperlactatemia
Record Dates: First submitted 2020-02-29; First posted 2020-03-19 (Actual); Last update posted 2020-03-19 (Actual); Status verified 2020-03

CONDITIONS: Continuous Renal Replacement Therapy; Hyperlactatemia; Bleeding
MeSH Terms: conditions — Hyperlactatemia; Hemorrhage

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Reginal citrate anticoagulation (Experimental): Patients accepted regional citrate anticoagulation for CRRT. Blood flow 120-220 ml/h. Sodium citrate (4%) infusion before the filter in order to maintain post-filter ionCa2+ level between 0.25 to 0.35 mmol/L. Calcium gluconate supplementary after the filter to maintain serum ionCa2+ level between 1.0 to 1.2 mmol/L. Adjusting the infusion rate of sodium citrate and blood flow according to pre- and post-filtration ionCa2+. Adjusting the infusion rate of calcium gluconate according to the serum ionCa2+ level.
  Interventions: Procedure: Regional citrate anticoagulation CRRT
- No-anticoagulation (Active Comparator): Patients accepted no-anticoagulation CRRT. Blood flow 200 ml/h. The replacement fluid was infused 50% predilution and 50% post-dilution.
  Interventions: Procedure: No-anticoagulation CRRT

INTERVENTIONS:
Procedure: Regional citrate anticoagulation CRRT — Regional citrate anticoagulation Sodium citrate (4%) infusion before the filter in order to maintain post-filter ionCa2+ level between 0.25 to 0.35 mmol/L. Calcium gluconate supplementary after the filter to maintain serum ionCa2+ level between 1.0 to 1.2 mmol/L.
  Arms: Reginal citrate anticoagulation
Procedure: No-anticoagulation CRRT — Patients accepted no-anticoagulation CRRT. Blood flow 200 ml/h. The replacement fluid was infused 50% predilution and 50% post-dilution.
  Arms: No-anticoagulation

SUMMARY:
The purpose of this single center, randomized, control, open-labeled study is to evaluate the effect and safety of RCA versus no anticoagulation for CRRT in hyperlactatemia patients with increased bleeding risk.

DETAILED DESCRIPTION:
For continuous renal replacement therapy (CRRT) patients with shock and muscle hypoperfusion, which characterised by tissue hypoxia and hyperlactatemia, the Kidney Disease Improving Global Outcomes (KIDIGO) guideline recommended no use of regional citrate anticoagulation (RCA) considering the potential increased citrate accumulation (CA) risk. In the condition of increased bleeding, no-anticoagulation was recommended for these patients. However, CRRT processed without anticoagulation was proved to be associated with shorter filter lifespan. Therefore, the purpose of this single center, randomized, control, open-labeled study is to evaluate the safety and efficacy of RCA versus no-anticoagulation for CRRT in hyperlactatemia patients with increased bleeding risk.

ELIGIBILITY:
Inclusion Criteria:

* Age≥16 years
* Hyperlactatemia (Lactic acid or serum lactate level > 2 mmol/L)
* Required CRRT
* Increased bleeding risk: PLT < 40 x 109, aPTT > 60 s, INR > 1.5, bleeding or active bleeding within 7 days, recent trauma or surgery (especially head trauma and neurosurgery), recent stroke, intracranial venous malformation or aneurysm, retinal hemorrhage, uncontrolled hypertension, and epidural catheter implantation.

Exclusion Criteria:

* Drugs (biguanide, linezolid, cyanide, etc.) and congenital metabolic disorders (glucose-6 phosphatase and 1,6 phosphofructosase deficiency) and mitochondrial damage caused hyperlactatemia.
* Receiving systemic anticoagulant treatment (heparin/lmol/warfarin/aspirin, etc.) within 24 hours.
* Critical patients with lactic acid ≥15mmol\L (with a mortality of 100%) were excluded
* Patients with APTT > 100S were excluded (retrospective data suggested that this type of patients received CRRT treatment should last for more than 24 hours)
* Patients who are pregnant or during lactation
* Severe liver failure: child-pugh score >10 (chronic severe liver failure), MELD score > 30 (acute severe liver failure), total bilirubin >51 mol/L
* Patients with internal fistula were treated with CRRT
* Unable to cooperate with treatment due to mental problems (such as depression and mental illness)
* CRRT with arteriovenous fistula, or the prescribed treatment time < 12 hours

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2020-03-30 (Estimated); Primary Completion 2022-03-01 (Estimated); Study Completion 2022-03-03 (Estimated)

PRIMARY OUTCOMES:
Filter failure | 72 hours
  TMP (transmembrane pressure) ≥ 300 mmHg, extracorporeal coagulation due to blood clots

SECONDARY OUTCOMES:
Serum Total Ca2+/ion Ca2+ level | 2, 6, 12, 20, 28, 36, 44, 52, 60, and 72 hours
  Serum Total Ca2+/ion Ca2+ level
Serum AST level | Every 24 hours up to 72 hours
  AST
Serum total bilirubin level | Every 24 hours up to 72 hours
  Total bilirubin
Serum citrate concentration | 2, 6, 12, 20, 28, 36, 44, 52, 60, and 72 hours
  Citrate concentration
Serum lactate level | 2, 6, 12, 20, 28, 36, 44, 52, 60, and 72 hours
  Serum lactate level
citrate accumulation | 72 hours
  Metabolic acidosis with an increased anion gap, decreasing ionized calcium, elevated total calcium and the calcium ratio (totCa/ionCa) > 2.5 were considered as citrate accumulation.
Hypocalcemia | 72 hours
  Ionized Ca2+ < 1.0
Acidosis | 72 hours
  Blood pH < 7.35
Alkalosis | 72 hours
  Blood pH > 7.45
Bleeding | 72 hours
  Bleeding episode during the CRRT
APTT | Every 24 hours up to 72 hours
  activated partial thromboplastin time
PT | Every 24 hours up to 72 hours
  Prothrombin time
INR | Every 24 hours up to 72 hours
  International normalized ratio
Mortality | Up to 3 months
  In-hospital mortality

CONTACTS AND LOCATIONS:
Overall Officials: Shiren Sun, MD, Principal Investigator — Xijing Hospital
Locations (1):
- Xijing Hospital of Nephrology, Xi'an, Shaanxi, China

IPD SHARING:
Plan to Share IPD: No